CLINICAL TRIAL: NCT03053180
Title: Real World Evidence Study of the Effectiveness of Paritaprevir/r - Ombitasvir, + Dasabuvir Without Ribavirin in Patients With Chronic HCV Gt1b Infection and Compensated Liver Cirrhosis in the RussIan FederaTion- An ObseRvational, MultI-CeNter Study (CITRIN)
Brief Title: Real World Evidence of the Effectiveness of Paritaprevir/Ritonavir (r) - Ombitasvir, + Dasabuvir Without Ribavirin in Participants With Chronic Hepatitis C and Compensated Liver Cirrhosis in the Russian Federation
Acronym: CITRIN
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-253
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Chronic Hepatitis C
Keywords: Paritaprevir; Dasabuvir; Ombitasvir; Ritonavir; Ribavirin free; Chronic Hepatitis C genotype 1b (GT1b); Cirrhosis; Compensated liver cirrhosis; Hepatitis
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir: Participants with chronic hepatitis C (CHC) genotype 1b (GT1b) and compensated liver cirrhosis received paritaprevir/ritonavir (r), ombitasvir and dasabuvir (3DAA ABBVIE REGIMEN) for 12 weeks.
  The prescription of a treatment regimen was at the discretion of the physician in accordance with local clinical practice and label, was made independently from this observational study and preceded the decision to offer a patient the opportunity to participate in this study.

SUMMARY:
This prospective, multi-center, observational study is designed to assess the real world effectiveness of paritaprevir/r - ombitasvir with dasabuvir (3DAA [direct-acting antiviral agent] ABBVIE REGIMEN) without ribavirin (RBV) and to describe baseline characteristics of participants with chronic hepatitis C virus (HCV) genotype 1b (GT1b) infection and compensated liver cirrhosis in Russia.

ELIGIBILITY:
Inclusion Criteria:

* 3DAA ABBVIE REGIMEN will be prescribed by physicians according to the routine clinical practice
* Treatment-naïve or interferon (IFN)/ribavirin (RBV)-experienced participants with confirmed CHC Gt1b and compensated liver cirrhosis, receiving therapy with the interferon-free 3DAA ABBVIE REGIMEN initiated not earlier than 2 weeks before the enrollment or the initiation is planned not later than 2 weeks after the day of enrollment in accordance to standard of care and in line with the current local label
* Participants must not be participating or intending to participate in a concurrent interventional therapeutic trial

Exclusion Criteria:

* Co-administration ribavirin (RBV) with the 3DAA ABBVIE REGIMEN
* Participants with Child Pugh B and C cirrhosis
* Participants with a history of prior direct-acting antiviral agent (DAA) therapy
* Any other contraindications to the administration of 3DAA ABBVIE REGIMEN according to the label

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic hepatitis C (CHC) genotype 1 (GT1b) and compensated liver cirrhosis will be recruited and observed in approximately 5-7 national and regional hospitals/outpatient services in Russia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (7):
- Russia (7):
  - South-Ural State Med. Academy, Chelyabinsk
  - KOGBUZ Kirovsk Infect Hosp, Kirov
  - Specialized Clinical Infectiou, Krasnodar
  - Orenburg Regional Clinical Hos, Orenburg
  - LLC Medical Company, Samara
  - GBOU VPO Saratov state Med Uni, Saratov
  - Ulyanovsk Regional Clin Hosp, Ulyanovsk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 participants signed the written patient authorization form and were enrolled into the study in 7 investigational sites located in Russia.
Groups:
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir: Participants with chronic hepatitis C (CHC) genotype 1b (GT1b) and compensated liver cirrhosis received paritaprevir/ritonavir (r), ombitasvir and dasabuvir (3 direct-acting antiviral agent [3DAA] ABBVIE REGIMEN) for 12 weeks.
  The prescription of a treatment regimen was at the discretion of the physician in accordance with local clinical practice and label, was made independently from this observational study and preceded the decision to offer a patient the opportunity to participate in this study.
Period: Overall Study
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
Started | 60
Completed | 59
Not Completed | 1
Not completed — Failure to Return | 1

BASELINE CHARACTERISTICS:
Population: The Core Population included all participants who had started and received the treatment combination recommended in the current local label for their disease characteristic and with end of treatment (EoT) > study day 55 (8 weeks).
Groups:
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir: Participants with chronic hepatitis C (CHC) genotype 1b (GT1b) and compensated liver cirrhosis received paritaprevir/ritonavir (r), ombitasvir and dasabuvir (3DAA ABBVIE REGIMEN) for 12 weeks.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) ribonucleic acid (RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last dose of study drug (week 24)
Population: Core population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
Number analyzed (Participants) | 59
percentage of participants | 98.3 [90.91 to 99.96]

2. Secondary Outcome: Percentage of Participants Achieving Virological Response at End of Treatment (EoT)
Description: Virological response is defined as HCV RNA less than 50 IU/mL.
Time Frame: End of treatment, maximum of 12 weeks
Population: Core population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
Number analyzed (Participants) | 59
percentage of participants | 100.0 [93.94 to 100.00]

3. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as participants with a virologic response (VR; HCV RNA < 50 IU/mL) at end of treatment (EOT) followed by HCV RNA ≥ 50 IU/mL at any time after the end of treatment.
Time Frame: End of treatment (week 12) and up to 12 weeks after the end of treatment.
Population: Core population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
Number analyzed (Participants) | 59
percentage of participants | 0.0 [0.00 to 6.06]

4. Secondary Outcome: Percentage of Participants With Breakthrough
Description: Breakthrough was defined as at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment.
Time Frame: 12 weeks
Population: Core population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
Number analyzed (Participants) | 59
percentage of participants | 0.0 [0.00 to 6.06]

5. Secondary Outcome: Percentage of Participants With Failure to Suppress
Description: Failure to suppress was defined as each measured on-treatment HCV RNA value ≥ 50 IU/mL.
Time Frame: 12 weeks
Population: Core population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
Number analyzed (Participants) | 59
percentage of participants | 0.0 [0.00 to 6.06]

6. Secondary Outcome: Percentage of Participants With Missing SVR12 Data
Time Frame: 12 weeks after the last dose of study drug (week 24)
Population: Core population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
Number analyzed (Participants) | 59
percentage of participants | 1.7 [0.04 to 9.09]

ADVERSE EVENTS:
Time Frame: From first dose of the 3DAA ABBVIE REGIMEN through 30 days after last dose (up to 16 weeks).
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 1/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir (N=60)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir (N=60)
Ascariasis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT03053180/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03053180/SAP_001.pdf